CLINICAL TRIAL: NCT02000115
Title: Portico Re-sheathable Transcatheter Aortic Valve System US IDE Trial
Acronym: PORTICO-IDE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1203
Record Dates: First submitted 2013-11-26; First posted 2013-12-03 (Estimated); Results first posted 2021-01-12 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Aortic Valve Stenosis
Keywords: Portico
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Randomized IDE Cohort, Portico Valve (Experimental): Portico transcatheter aortic valve and Portico delivery system.
  Status: ACTIVE, NOT ENROLLING.
  Interventions: Device: Portico transcatheter aortic valve
- Randomized IDE Cohort, CAV (Active Comparator): Any FDA approved, commercially-available transcatheter aortic valve (CAV).
  Status: ACTIVE, NOT ENROLLING.
  Interventions: Device: Commercially available transcatheter aortic valve
- Nested Valve-in-Valve Registry (Experimental): Subjects who have documented failed aortic surgical valve prosthesis and are deemed eligible to receive a transcatheter Portico valve
  Status: ACTIVE, ENROLLING.
  Interventions: Device: Portico transcatheter aortic valve
- FlexNav Delivery System Study (Experimental): Portico transcatheter aortic valve and FlexNav delivery system
  Status: ACTIVE, NOT ENROLLING
  Interventions: Device: Portico transcatheter aortic valve

INTERVENTIONS:
Device: Portico transcatheter aortic valve — St. Jude Medical transcatheter Portico aortic valve
  Arms: FlexNav Delivery System Study; Nested Valve-in-Valve Registry; Randomized IDE Cohort, Portico Valve
Device: Commercially available transcatheter aortic valve — Commercially available transcatheter aortic valve
  Arms: Randomized IDE Cohort, CAV

SUMMARY:
The objective of the PORTICO pivotal IDE trial is to evaluate the safety and effectiveness of the St Jude Medical (SJM) Portico Transcatheter Heart Valve and Delivery Systems (Portico) in the treatment of severe symptomatic aortic stenosis via transfemoral and alternative delivery methods in high risk and extreme risk patients.

DETAILED DESCRIPTION:
The PORTICO pivotal IDE trial will include a randomized cohort of 750 subjects enrolled at up to 70 investigational sites in the United States and Australia. Patients will be randomized (1:1) to receive the SJM Portico Transcatheter Heart Valve and Delivery Systems (Portico) or any FDA-approved, commercially-available Transcatheter Aortic Valve Replacement (TAVR) System. The randomized cohort will be tested for two co-primary endpoints at 30 days (primary safety endpoint) and 1 year (primary effectiveness endpoint). At the time of the primary randomized cohort analysis, the risk cohorts will be combined and analysis will be conducted on the intention-to-treat (n=750) population.

The FlexNav Delivery System study will be conducted as a separate arm of the PORTICO IDE trial and will include up to 200 high or extreme risk subjects; including a minimum of 100 analysis subjects. The study will characterize the safety of the next-generation Portico Delivery System ("FlexNav™ Delivery System"). The primary analysis cohort will include FlexNav analysis subjects.

The IDE Valve-in-Valve registry will enroll up to 100 high or extreme risk subjects with a failed surgical bioprosthesis who are eligible to receive a Portico Transcatheter Heart Valve.

All subjects enrolled in the PORTICO pivotal IDE trial will undergo follow-up at baseline, peri- and post-procedure, at discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, 12-months and then annually through 5-years.

ELIGIBILITY:
Inclusion Criteria

1. Subjects must have co-morbidities such that the surgeon and cardiologist Co-Investigators concur that the predicted risk of operative mortality is ≥15% or a minimum Society of Thoracic Surgeons (STS) score of 8%. A candidate who does not meet the STS score criteria of ≥ 8% can be included in the study if a peer review by at least two surgeons concludes and documents that the patient's predicted risk of operative mortality is ≥15%. The surgeon's assessment of operative comorbidities not captured by the STS score must be documented in the study case report form as well as in the patient medical record.
2. Subject is 21 years of age or older at the time of consent.
3. Subject has senile degenerative aortic valve stenosis with echocardiographically derived criteria: mean gradient >40 mmHg or jet velocity greater than 4.0 m/s or Doppler Velocity Index <0.25 and an initial aortic valve area (AVA) of ≤ 1.0 cm2 (indexed effective orifice area (EOA) ≤ 0.6 cm2/m2). (Qualifying AVA baseline measurement must be within 60 days prior to informed consent).
4. Subject has symptomatic aortic stenosis as demonstrated by New York Heart Association (NYHA) Functional Classification of II, III, or IV.
5. The subject has been informed of the nature of the study, agrees to its provisions and has provided written informed consent as approved by the Institutional Review Board (IRB) of the respective clinical site.
6. The subject and the treating physician agree that the subject will return for all required post-procedure follow-up visits.
7. Subject's aortic annulus is 19-27mm diameter as measured by computerized tomography (CT) conducted within 12 months prior to informed consent. Note: if CT is contraindicated and/or not possible to be obtained for certain subjects, a 3D echo and non-contrast CT of chest and abdomen/pelvis may be accepted if approved by the subject selection committee.

   For a subject to be considered an Extreme Risk candidate they must meet # 2, 3, 4, 5, 6, 7 of the above criteria, and
8. The subject, after formal consults by a cardiologist and two cardiovascular surgeons agree that medical factors preclude operation, based on a conclusion that the probability of death or serious, irreversible morbidity exceeds the probability of meaningful improvement. Specifically, the probability of death or serious, irreversible morbidity should exceed 50%. The surgeons' consult notes shall specify the medical or anatomic factors leading to that conclusion and include a printout of the calculation of the STS score to additionally identify the risks in these patients.

Exclusion Criteria

1. Evidence of an acute myocardial infarction (defined as: ST Segment Elevation as evidenced on 12 Lead ECG) within 30 days prior to index procedure.
2. Aortic valve is a congenital unicuspid or congenital bicuspid valve or is non-calcified as verified by echocardiography.
3. Mixed aortic valve disease (aortic stenosis and aortic regurgitation with predominant aortic regurgitation 3-4+).
4. Any percutaneous coronary or peripheral interventional procedure performed within 30 days prior to index procedure.
5. Pre-existing prosthetic heart valve or other implant in any valve position, prosthetic ring, severe circumferential mitral annular calcification (MAC) which is continuous with calcium in the left ventricular outflow tract (LVOT), severe (greater than 3+) mitral insufficiency, or severe mitral stenosis with pulmonary compromise. Subjects with pre-existing surgical bioprosthetic aortic heart valve should be considered for the Valve-in-Valve registry.
6. Blood dyscrasias as defined: leukopenia (WBC<3000 mm3), acute anemia (Hb < 9 g/dL), thrombocytopenia (platelet count <50,000 cells/mm³).
7. History of bleeding diathesis or coagulopathy.
8. Cardiogenic shock manifested by low cardiac output, vasopressor dependence, or mechanical hemodynamic support.
9. Untreated clinically significant coronary artery disease requiring revascularization.
10. Hemodynamic instability requiring inotropic support or mechanical heart assistance.
11. Need for emergency surgery for any reason.
12. Hypertrophic cardiomyopathy with or without obstruction (HOCM).
13. Severe ventricular dysfunction with left ventricular ejection fraction (LVEF) <20% as measured by resting echocardiogram.
14. Echocardiographic evidence of intracardiac mass, thrombus or vegetation.
15. Active peptic ulcer or upper gastrointestinal (GI) bleeding within 3 months prior to index procedure.
16. A known hypersensitivity or contraindication to aspirin, heparin, ticlopidine (Ticlid), or clopidogrel (Plavix), or sensitivity to contrast media which cannot be adequately premedicated.
17. Recent (within 6 months prior to index procedure date) cerebrovascular accident (CVA) or a transient ischemic attack (TIA).
18. Renal insufficiency (creatinine > 3.0 mg/dL) and/or end stage renal disease requiring chronic dialysis.
19. Life expectancy < 12 months from the time of informed consent due to non-cardiac co-morbid conditions.
20. Significant aortic disease, including abdominal aortic or thoracic aneurysm defined as maximal luminal diameter 5cm or greater; marked tortuosity (hyperacute bend), aortic arch atheroma (especially if thick [> 5 mm], protruding or ulcerated) or narrowing (especially with calcification and surface irregularities) of the abdominal or thoracic aorta, severe "unfolding" and tortuosity of the thoracic aorta (applicable for transfemoral patients only).
21. Native aortic annulus size < 19 mm or > 27 mm per the baseline diagnostic imaging.
22. Aortic root angulation > 70° (applicable for transfemoral patients only).
23. Currently participating in an investigational drug or device study.
24. Active bacterial endocarditis within 6 months prior to the index procedure.
25. Bulky calcified aortic valve leaflets in close proximity to coronary ostia.
26. Non-calcified aortic annulus
27. Iliofemoral vessel characteristics that would preclude safe placement of the introducer sheath such as severe obstructive calcification, or severe tortuosity (applicable for transfemoral patients only).

Additional Exclusion Criteria (Transcatheter Access Related)

For selection of an appropriate alternative access delivery method, subjects were screened using the following access specific exclusion criteria:

Transaortic (TAo) Subject Cohort Specific Exclusion Criteria

1. Subject has pre-existing patent RIMA graft that would preclude access.
2. Subject has a hostile chest or other condition that complicates transaortic access.
3. Subject has a porcelain aorta, defined as an extensive circumferential calcification of the ascending aorta that would complicate TAo access.

Additional exclusion criteria for transaortic access using the FlexNav™ Delivery System:

1. Subject has a distance between the annular plane and the aortic access site <7 cm (2.8")
2. Subject has a distance between the annular plane and the separate introducer sheath distal tip <6 cm (2.4")

Subclavian/Axillary Subject Cohort Specific Exclusion Criteria

1. Subject's access vessel (subclavian/axillary) diameter will not allow for introduction of the applicable 18 Fr or 19 Fr delivery system.
2. Subject's subclavian/axillary arteries have severe calcification and/or tortuosity.
3. Subject's aortic root angulation is:

   * Left Subclavian/Left Axillary: >70◦
   * Right Subclavian/Right Axillary: >30◦
4. Subject has a history of patent LIMA/RIMA graft that would preclude access

Additional exclusion criteria for subclavian/axillary access using the FlexNav™ Delivery System:

1. Subject's access vessel (subclavian/axillary) has a distance between the annular plane and the integrated sheath distal tip <17 cm (6.7")
2. Subject's access vessel requires the delivery system to be advanced through a separate introducer sheath

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1242 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2026-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Raj R Makkar, MD, Principal Investigator — Cedars-Sinai Medical Center; Gregory P Fontana, MD, Principal Investigator — Los Robles Regional Medical Center
Locations (70):
- United States (65):
  - University Hospital - Univ. of Alabama at Birmingham (UAB), Birmingham, Alabama
  - Banner - University Medical Center Phoenix, Phoenix, Arizona
  - John Muir Medical Center, Concord, California
  - Scripps Green Hospital, La Jolla, California
  - USC University Hospital, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Stanford University Medical Center, Palo Alto, California
  - Huntington Memorial Hospital, Pasadena, California
  - Sutter Memorial Hospital, Sacramento, California
  - Mercy General Hospital, Sacramento, California
  - Los Robles Regional Medical Center, Thousand Oaks, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - JFK Medical Center, Atlantis, Florida
  - Morton Plant Valve Clinic, Clearwater, Florida
  - Delray Medical Center, Delray Beach, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - St. Vincent Hospital, Indianapolis, Indiana
  - Iowa Heart Center, West Des Moines, Iowa
  - Cardiovascular Research Institute of Kansas, Wichita, Kansas
  - Ochsner Medical Center, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - North Mississippi Medical Center, Tupelo, Mississippi
  - St. Luke's Hospital, Kansas City, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Catholic Medical Center, Manchester, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Albany Medical Center, Albany, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Winthrop University Hospital, Mineola, New York
  - New York Presbyterian Hospital / Cornell University, New York, New York
  - Lenox Hill Hospital, New York, New York
  - St. Francis Hospital, Roslyn, New York
  - Mission Health and Hospitals, Asheville, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina Heart Institute, Greenville, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - Pinnacle Health System, Harrisburg, Pennsylvania
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny Singer Research Institute, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Main Line Health Center/Lankenau Hospital, Wynnewood, Pennsylvania
  - Sanford USD Medical Center, Sioux Falls, South Dakota
  - Baptist Memorial Hospital, Memphis, Tennessee
  - Centennial Medical Center, Nashville, Tennessee
  - Heart Hospital of Austin, Austin, Texas
  - CHI St. Luke's Health Baylor College of Medicine Medical Center, Houston, Texas
  - Memorial Hermann Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Swedish Medical Center, Seattle, Washington
- Australia (5):
  - Macquarie University Hospital, Sydney, New South Wales
  - The Prince Charles Hospital, Chermside, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia

REFERENCES:
- [Derived] Puri R, Thiele H, Fichtlscherer S, Westermann D, Makkar R, Waksman R, Hakmi S, Sondergaard L, Groh M, Montarello JK, Kempfert J, Yong G, Bedogni F, Maisano F, Worthley SG, Rodes-Cabau J, Fontana GP, Mollmann H. Five-Year Clinical Outcomes and Durability of a Self-Expanding Transcatheter Heart Valve With Intra-Annular Leaflets. Circ Cardiovasc Interv. 2025 Dec;18(12):e015430. doi: 10.1161/CIRCINTERVENTIONS.125.015430. Epub 2025 Oct 24. PMID 41133305
- [Derived] Makkar RR, Cheng W, Waksman R, Satler LF, Chakravarty T, Groh M, Abernethy W, Russo MJ, Heimansohn D, Hermiller J, Worthley S, Chehab B, Cunningham M, Matthews R, Ramana RK, Yong G, Ruiz CE, Chen C, Asch FM, Nakamura M, Jilaihawi H, Sharma R, Yoon SH, Pichard AD, Kapadia S, Reardon MJ, Bhatt DL, Fontana GP. Self-expanding intra-annular versus commercially available transcatheter heart valves in high and extreme risk patients with severe aortic stenosis (PORTICO IDE): a randomised, controlled, non-inferiority trial. Lancet. 2020 Sep 5;396(10252):669-683. doi: 10.1016/S0140-6736(20)31358-1. Epub 2020 Jun 25. PMID 32593323
- [Derived] Makkar RR, Fontana G, Jilaihawi H, Chakravarty T, Kofoed KF, De Backer O, Asch FM, Ruiz CE, Olsen NT, Trento A, Friedman J, Berman D, Cheng W, Kashif M, Jelnin V, Kliger CA, Guo H, Pichard AD, Weissman NJ, Kapadia S, Manasse E, Bhatt DL, Leon MB, Sondergaard L. Possible Subclinical Leaflet Thrombosis in Bioprosthetic Aortic Valves. N Engl J Med. 2015 Nov 19;373(21):2015-24. doi: 10.1056/NEJMoa1509233. Epub 2015 Oct 5. PMID 26436963

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 750 subjects were randomized (1:1) to the Portico valve (n=381) and CAV (n=369) groups.
  100 analysis subjects were enrolled in the FlexNav Delivery System study.
  53 subjects are currently enrolled in the IDE Valve-in-Valve registry ( enrollment ongoing)
Pre-assignment Details: Only the Randomized IDE cohort (N=750) and FlexNav Delivery System Study (N=100 analysis) that completed subject enrollment and reached their pre-defined primary endpoint(s) are included in the Results Section.
  The IDE Valve-in-Valve registry is still enrolling subjects. A total of 53 out of a required 100 subjects have been enrolled to date.
Groups:
- Randomized IDE Cohort, Portico Valve: Portico transcatheter aortic valve and Portico delivery System.
- Randomized IDE Cohort, CAV: Any FDA approved, commercially-available transcatheter aortic valve (CAV).
- FlexNav Delivery System Study: Portico transcatheter aortic valve and FlexNav delivery system
- Nested Valve-in-Valve Registry: Subjects who have documented failed aortic surgical valve prosthesis and are deemed eligible to receive a transcatheter Portico valve
Period: Overall Study
Arm/Group | Randomized IDE Cohort, Portico Valve | Randomized IDE Cohort, CAV | FlexNav Delivery System Study | Nested Valve-in-Valve Registry
Started | 381 | 369 | 100 | 53
Completed | 302 (6 subjects missed the One-year follow-up visit) | 301 (8 subjects missed the One-year follow-up visit) | 99 (1 subject missed the 30 day follow-up visit) | 0
Not Completed | 79 | 68 | 1 | 53
Not completed — Death | 56 | 45 | 0 | 0
Not completed — Missed Visit | 6 | 8 | 1 | 0
Not completed — Protocol Violation | 2 | 1 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 11 | 11 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Non-compliance | 2 | 1 | 0 | 0
Not completed — Withdrawn on day of randomization | 0 | 1 | 0 | 0
Not completed — Still on Study | 0 | 0 | 0 | 53

BASELINE CHARACTERISTICS:
Population: Randomized IDE cohort: analysis population includes all randomized subjects (intention-to-treat) FlexNav Delivery System study: analysis population includes all enrolled subjects (defined as insertion of FlexNav delivery system into subject's vasculature)
Groups:
- Total: Total of all reporting groups
Arm/Group | Randomized IDE Cohort, Portico Valve | Randomized IDE Cohort, CAV | FlexNav Delivery System Study | Total
Number analyzed (Participants) | 381 | 369 | 100 | 850
Age, Continuous [Mean (Standard Deviation); unit: years] | 83.0 (7.6) | 83.7 (7.0) | 85.1 (5.8) | 83.5 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 198 | 197 | 57 | 452
  Male | 183 | 172 | 43 | 398
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 354 | 339 | 92 | 785
  Race: Black or African American | 14 | 17 | 7 | 38
  Race: American Indian or Alaska native | 1 | 0 | 1 | 2
  Race: Asian | 4 | 3 | 0 | 7
  Race: Native Hawaiian or other Pacific Islander | 1 | 1 | 0 | 2
  Race: Other | 7 | 9 | 0 | 16
  Race: Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 351 | 340 | 75 | 796
  Australia | 30 | 29 | 25 | 88

OUTCOME MEASURES:

1. Primary Outcome: Primary Effectiveness Endpoint (Randomized IDE Cohort)
Description: A composite of all-cause mortality or disabling stroke at one year.
Time Frame: One-year from randomization
Population: Intention-to-treat analysis population.
Measure: Mean (Standard Error); unit: percentage of participants
Arm/Group | Randomized IDE Cohort, Portico Valve | Randomized IDE Cohort, CAV
Number analyzed (Participants) | 381 | 369
percentage of participants | 14.8 (1.8) | 13.4 (1.8)
Statistical Analysis 1: Comparison: Randomized IDE Cohort, Portico Valve vs Randomized IDE Cohort, CAV; We analysed the primary effectiveness endpoint in the intention-to- treat (ITT) population using the Kaplan-Meier method to estimate event rates, the Greenwood method to calculate the standard error of the Kaplan-Meier estimates, and assuming an asymptotic normal distribution for event rate estimates; Test type: Non-Inferiority — 8.0% non-inferiority margin; p = 0.006, Kaplan-Meier estimates — p for non-inferiority; Kaplan-Meier was used as the method for calculating the endpoint rate; Difference in percentages between groups = 1.5, 95% CI 1-sided [upper limit 5.7] — Non-inferiority of the Portico valve to commercially available valves was shown if the upper bound of the 95% confidence interval (1-sided) for the difference in event rates between groups was less than the non-inferiority margin (8·0%)

2. Primary Outcome: Primary Safety Endpoint (Randomized IDE Cohort)
Description: Non-hierarchical composite of all-cause mortality, disabling stroke, life threatening bleeding requiring blood transfusion, acute kidney injury requiring dialysis, or major vascular complications at 30 days.
Time Frame: 30 days from randomization
Population: Intention-to-treat analysis population
Measure: Mean (Standard Deviation); unit: percentage of participants
Arm/Group | Randomized IDE Cohort, Portico Valve | Randomized IDE Cohort, CAV
Number analyzed (Participants) | 381 | 369
percentage of participants | 13.8 (1.8) | 9.6 (1.5)
Statistical Analysis 1: Comparison: Randomized IDE Cohort, Portico Valve vs Randomized IDE Cohort, CAV; We analysed the primary safety endpoint in the intention-to-treat (ITT) population using the Kaplan-Meier method to estimate event rates, the Greenwood method to calculate the standard error of the Kaplan-Meier estimates, and assuming an asymptotic normal distribution for event rate estimates; Test type: Non-Inferiority — 8.5% non-inferiority margin; p = 0.03, Kaplan-Meier estimates — p for non-inferiority; Kaplan-Meier was used as the method for calculating the endpoint rate; Difference in percentages between groups = 4.2, 95% CI 1-sided [upper limit 8.1] — Non-inferiority of the Portico valve to commercially available valves was shown if the upper bound of the 95% confidence interval (1-sided) for the difference in event rates between groups was less than the non-inferiority margin (8·5%)

3. Primary Outcome: Percentage of Patients With Major Vascular Complications (Primary Safety Endpoint- FlexNav Delivery System Study)
Description: Valve Academic Research Consortium (VARC) 2- defined major vascular complications
Time Frame: 30 days from index procedure
Population: All enrolled analysis subjects
Measure: Number; unit: percentage of participants
Arm/Group | FlexNav Delivery System Study
Number analyzed (Participants) | 100
percentage of participants | 6.0

4. Secondary Outcome: Percentage of Patients With Severe Aortic Regurgitation (Randomized IDE Cohort)
Description: Severe aortic regurgitation (AR) at one year
Time Frame: One year
Population: All randomized subjects with available data at one-year
Measure: Number; unit: percentage of participants
Arm/Group | Randomized IDE Cohort, Portico Valve | Randomized IDE Cohort, CAV
Number analyzed (Participants) | 269 | 269
percentage of participants | 0.4 | 0
Statistical Analysis 1: Comparison: Randomized IDE Cohort, Portico Valve vs Randomized IDE Cohort, CAV; Test type: Non-Inferiority — non-inferiority margin of 4%; p = 0.001, Farrington-Manning test — p for non-inferiority; The test statistic is based on the Farrington-Manning method of testing non-inferiority of proportions; Difference in percentages between groups = 0.4, 95% CI 1-sided [upper limit 2.3] — If the upper limit of the 95% confidence interval (1-sided) for the difference of proportions (Portico - CAV) is < 4%, then non inferiority is demonstrated

5. Secondary Outcome: Kansas City Cardiomyopathy Questionnaire (KCCQ) Overall Summary Score (Randomized IDE Cohort)
Description: Kansas City Cardiomyopathy Questionnaire (KCCQ) at one year. Scale 0 to 100; with higher scores indicating better symptoms and physical functioning
Time Frame: One year
Population: All randomized subjects with available data at one-year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Randomized IDE Cohort, Portico Valve | Randomized IDE Cohort, CAV
Number analyzed (Participants) | 274 | 283
units on a scale | 75.4 (22.2) | 75.9 (20.5)
Statistical Analysis 1: Comparison: Randomized IDE Cohort, Portico Valve vs Randomized IDE Cohort, CAV; Test type: Non-Inferiority — non-inferiority margin of 10 points; p < 0.0001, two-sample t-test — p for non-inferiority; The test statistic is based on two sample t-test; Mean Difference (Final Values) = -0.5, 95% CI 1-sided [lower limit -3.5] — If the lower limit of the 95% confidence interval (1-sided) for the difference of (Portico - CAV) is > -10, then non inferiority is demonstrated

6. Secondary Outcome: Percentage of Patients With Moderate or Severe Aortic Regurgitation (Randomized IDE Cohort)
Description: Moderate or severe aortic regurgitation at one year
Time Frame: One year
Population: All randomized subjects with available data at one-year
Measure: Number; unit: percentage of participants
Arm/Group | Randomized IDE Cohort, Portico Valve | Randomized IDE Cohort, CAV
Number analyzed (Participants) | 269 | 269
percentage of participants | 7.1 | 1.5
Statistical Analysis 1: Comparison: Randomized IDE Cohort, Portico Valve vs Randomized IDE Cohort, CAV; Test type: Non-Inferiority — non-inferiority margin of 6%; p = 0.40, Farrington-Manning test — p for non-inferiority; The test statistic is based on the Farrington-Manning method of testing non-inferiority of proportions; Difference in percentages between groups = 5.6, 95% CI 1-sided [upper limit 8.5] — If the upper limit of the 95% confidence interval (1-sided) for the difference of proportions (Portico - CAV) is < 6%, then non inferiority is demonstrated

7. Secondary Outcome: Six-Minute Walk Test- Total Distance Walked (Randomized IDE Cohort)
Description: Six-minute walk distance at one year
Time Frame: One year
Population: All randomized subjects with available data at one-year
Measure: Mean (Standard Deviation); unit: meters
Groups:
- Randomized IDE Cohort, CAV: Any FDA approved, commercially-available transcatheter aortic valve (CAV).
  Status: ACTIVE, NOT ENROLLING.
  Commercially available transcatheter aortic valve: Commercially available transcatheter aortic valve
Arm/Group | Randomized IDE Cohort, Portico Valve | Randomized IDE Cohort, CAV
Number analyzed (Participants) | 227 | 225
meters | 235.0 (125.0) | 231.5 (118.5)
Statistical Analysis 1: Comparison: Randomized IDE Cohort, Portico Valve vs Randomized IDE Cohort, CAV; Test type: Non-Inferiority — non-inferiority margin on -36 meters; p = 0.0003, two sample t-test — p for non-inferiority; The test statistic is based on a two-sample t-test; Mean Difference (Final Values) = 3.5, 95% CI 1-sided [lower limit -15.4] — If the lower limit of the 95% confidence interval (1-sided) for the difference of (Portico - CAV) is > -36, then non inferiority is demonstrated

8. Secondary Outcome: Percentage of Patients With Composite Safety Endpoint (Nested Valve-in-Valve Registry)
Description: Non-hierarchical composite of all-cause mortality, disabling stroke, life threatening bleeding requiring blood transfusion, acute kidney injury requiring dialysis, or major vascular complications at 30 days from index procedure.
  Anticipated completion date (2022)
Time Frame: 30 days from index procedure
Reporting Status: Not Posted, anticipated posting 2026-12

9. Secondary Outcome: Percentage of Patients With All-cause Mortality or Disabling Stroke (Nested Valve-in-Valve Registry)
Description: A composite of all-cause mortality or disabling stroke at one year Anticipated completion data (2023)
Time Frame: One year from index procedure
Reporting Status: Not Posted, anticipated posting 2026-12

ADVERSE EVENTS:
Time Frame: Randomized IDE cohort: data reflects all serious and other (non serious) adverse events through 1 year in the intention-to-treat population (i.e. within 365 days of randomization); and all-cause mortality reflects all deaths through 1 year. FlexNav Delivery System study: data reflects all serious and other (non serious) adverse events through 30 days in the enrolled analysis population (i.e. within 30 days from index procedure); and all-cause mortality reflects all deaths through 30 days
Description: Site-reported Serious and Other (Not Including Serious) Adverse Events reflect data collected from the intention-to-treat population (RCT) or enrolled analysis population (FlexNav Delivery System Study); while All-Cause Mortality reflects the entire population
Arm/Group | Randomized IDE Cohort, Portico Valve | Randomized IDE Cohort, CAV | FlexNav Delivery System Study
All-Cause Mortality (participants affected / at risk) | 56/381 | 45/369 | 0/100
Serious Adverse Events (participants affected / at risk) | 273/381 | 231/369 | 44/100
Other Adverse Events (participants affected / at risk) | 298/381 | 269/369 | 54/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized IDE Cohort, Portico Valve (N=381) | Randomized IDE Cohort, CAV (N=369) | FlexNav Delivery System Study (N=100)
Angina Pectoris (Cardiac disorders) | 11 (14) | 6 (8) | 0 (0)
Aorta- Aortic Calcification (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic- Aortic Dissection (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Arrhythmias (Cardiac disorders) | 38 (43) | 34 (42) | 4 (4)
Arterial Hypertension (Cardiac disorders) | 3 (3) | 7 (7) | 0 (0)
EKG Abnormalities (Cardiac disorders) | 2 (2) | 3 (3) | 0 (0)
Echo finding (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Endocarditis- Infective/Bacterial Endocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Endocarditis- Prosthetic Valvular Endocarditis (PVE) (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
General- Asystole (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
General-Cardiac Arrest (Cardiac disorders) | 11 (12) | 3 (3) | 0 (0)
General- Cardiac Perforation (Cardiac disorders) | 4 (4) | 1 (1) | 0 (0)
General-Cardiomyopathy (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
General- Coronary Artery Disease (Cardiac disorders) | 2 (3) | 0 (0) | 1 (1)
General-Coronary Artery Occlusion (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
General-Hypertensive Crisis (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
General-Hypervolemia (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
General- Myocardial Ischemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
General- Pericardial Effusion (Cardiac disorders) | 7 (7) | 4 (4) | 0 (0)
General- Pericardial Tamponade (Cardiac disorders) | 7 (7) | 2 (2) | 2 (2)
General-Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
General-Pulmonary Hypertension (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
General- Cardiovascular Symptoms (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Heart Block (Cardiac disorders) | 98 (102) | 37 (39) | 12 (12)
Heart Failure (Cardiac disorders) | 56 (79) | 39 (52) | 3 (3)
Hypotension (Cardiac disorders) | 9 (9) | 3 (3) | 7 (7)
Myocardial Infarction (Cardiac disorders) | 7 (7) | 6 (6) | 0 (0)
Shock (Cardiac disorders) | 6 (6) | 6 (6) | 0 (0)
Valve- Aortic Valve Regurgitation/Aortic Valve Insufficiency/Valvular Regurgitation (Cardiac disorders) | 4 (4) | 1 (1) | 1 (1)
Valve- Aortic Valve Stenosis (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Valve- Mitral Valve Regurgitation/Mitral Insufficiency (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Valve- Mitral Valve Stenosis (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Valve- Perivalvular Leak (Cardiac disorders) | 13 (13) | 6 (6) | 0 (0)
Valve- Tricuspid Regurgitation/Tricuspid Insufficiency/Valvular Regurgitation Tricuspid Valve (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (5) | 0 (0)
General-Dematological (Skin and subcutaneous tissue disorders) | 4 (5) | 6 (7) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0)
Nose and Paranasal Sinuses (General disorders) | 1 (1) | 3 (3) | 0 (0)
Throat- Cough (General disorders) | 0 (0) | 1 (1) | 0 (0)
Disorders of Carbohydrate Metabolism (Metabolism and nutrition disorders) | 14 (16) | 11 (13) | 0 (0)
General- Fluid, Electrolyte, Endocine and Metabolic Disorders (Metabolism and nutrition disorders) | 14 (15) | 9 (10) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 3 (5) | 0 (0) | 0 (0)
Esophageal Laceration and Rupture (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
General-Gastrointestinal Disorders (Gastrointestinal disorders) | 31 (36) | 25 (26) | 3 (3)
General-Gastrointestinal Symptoms (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Hepatic and Biliary Disorders (Gastrointestinal disorders) | 3 (4) | 3 (4) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
General-Genitourinary Disorders (Renal and urinary disorders) | 21 (22) | 17 (19) | 2 (2)
General-Genitourinary Symptoms (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0)
Prostate Disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal Failure (Renal and urinary disorders) | 11 (11) | 9 (9) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 9 (9) | 14 (14) | 3 (3)
Breast Cancer (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Anemias (Blood and lymphatic system disorders) | 36 (37) | 32 (35) | 4 (4)
General-Hematology and Oncology (Blood and lymphatic system disorders) | 43 (48) | 21 (29) | 13 (18)
Fungal Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
General- Infections (Infections and infestations) | 14 (16) | 14 (14) | 1 (1)
Allergy (General disorders) | 2 (2) | 0 (0) | 0 (0)
Miscellaneous- Device Malposition or Malfunction (Product Issues) | 3 (3) | 2 (2) | 0 (0)
Miscellaneous- Device Migration (Product Issues) | 1 (1) | 0 (0) | 2 (2)
Miscellaneous-Thrombus on Device (Product Issues) | 5 (5) | 1 (1) | 0 (0)
Miscellaneous- General (General disorders) | 60 (68) | 60 (70) | 4 (5)
Fracture (Musculoskeletal and connective tissue disorders) | 11 (11) | 11 (11) | 1 (1)
General-Musculoskeletal and Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 0 (0)
General- Musculoskeletal Symptoms (Musculoskeletal and connective tissue disorders) | 8 (9) | 3 (4) | 0 (0)
Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
General-Neurological (Nervous system disorders) | 33 (34) | 18 (25) | 5 (5)
General- Neurological Symptoms (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0)
Hemorrhage (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0)
Neurological Hematoma (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Seizure/Convulsions/Epilepsy (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0)
Stroke (Nervous system disorders) | 11 (11) | 18 (20) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 1 (1)
Chronic Obstructive Airway Disorders (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (8) | 1 (1)
General- Pulmonary/Respiratory Disorders (Respiratory, thoracic and mediastinal disorders) | 36 (48) | 26 (28) | 3 (3)
Eosinophilic Pneumonias (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0)
Idiopathic Interstitial Lung Diseases (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural Disorders (Respiratory, thoracic and mediastinal disorders) | 12 (14) | 9 (9) | 3 (3)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 26 (29) | 16 (16) | 2 (2)
VASC Bleeding (Injury, poisoning and procedural complications) | 4 (4) | 2 (2) | 2 (2)
VASC Hematoma (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
VASC Pseudoaneurysm (Injury, poisoning and procedural complications) | 8 (8) | 4 (4) | 1 (1)
VASC Vascular Rupture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
VASC Vessel Dissection (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
VASC Vessel Perforation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
VASC Vessel Stenosis (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Hypovolemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized IDE Cohort, Portico Valve (N=381) | Randomized IDE Cohort, CAV (N=369) | FlexNav Delivery System Study (N=100)
Angina Pectoris (Cardiac disorders) | 11 (12) | 9 (9) | 1 (1)
Aortic-Aortic Dissection (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0)
Arrhythmias (Cardiac disorders) | 54 (60) | 45 (50) | 11 (11)
Arterial Hypertension (Cardiac disorders) | 19 (19) | 10 (10) | 1 (1)
EKG Abnormalities (Cardiac disorders) | 3 (3) | 4 (4) | 0 (0)
Echo Finding (Cardiac disorders) | 2 (2) | 5 (5) | 0 (0)
General (Cardiac disorders) | 23 (23) | 19 (20) | 8 (8)
General- Cardiovascular Symptoms (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Heart Block (Cardiac disorders) | 102 (114) | 83 (91) | 19 (20)
Heart Failure (Cardiac disorders) | 22 (23) | 22 (22) | 1 (1)
Hypotension (Cardiac disorders) | 15 (15) | 11 (11) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Valve-Aortic Valve Regurgitation/Aortic Valve Insufficiency/Valvular Regurgitation Aortic Valve (Cardiac disorders) | 16 (16) | 5 (5) | 4 (4)
Valve- Aortic Valve Stenosis (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Valve- Mitral Valve Regurgitation/Mitral Insufficiency (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0)
Valve- Perivalvular Leak (Cardiac disorders) | 21 (21) | 8 (8) | 2 (2)
Valve-Tricuspid Regurgitation/Tricuspid Insufficiency/Valvular Regurgitation Tricuspid Valve (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Cardiomegaly (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (5) | 0 (0)
General-Dermatogical (Skin and subcutaneous tissue disorders) | 6 (6) | 11 (12) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 4 (4) | 3 (3) | 0 (0)
Dental Disorders (General disorders) | 3 (3) | 2 (2) | 0 (0)
Nose and Paranasal Sinuses (General disorders) | 7 (8) | 2 (2) | 0 (0)
Throat (General disorders) | 1 (1) | 3 (3) | 0 (0)
Disorders of Carbohydrate Metabolism (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 0 (0)
General- Fluid, Electrolyte, Endocrine and Metabolic Disorders (Metabolism and nutrition disorders) | 26 (34) | 18 (22) | 2 (2)
Thyroid Disorders (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Esophageal Disorders (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
General (Gastrointestinal disorders) | 10 (13) | 10 (11) | 0 (0)
General- Gastrointestinal Symptoms (Gastrointestinal disorders) | 4 (5) | 1 (1) | 0 (0)
Hepatic and Biliary Disorders (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
General- Genitourinary Disorders (Renal and urinary disorders) | 35 (40) | 41 (42) | 6 (6)
General- Genitourinary Symptoms (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0)
Myoneurogenic Disorders (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Prostate Disease (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 3 (3) | 1 (1) | 0 (0)
Urinary Tract Infections (Renal and urinary disorders) | 33 (36) | 20 (21) | 1 (1)
Anemias (Blood and lymphatic system disorders) | 46 (48) | 40 (40) | 11 (11)
General- Hematology and Oncology (Blood and lymphatic system disorders) | 87 (105) | 56 (65) | 17 (18)
Fungal Infections (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
General- Infections (Infections and infestations) | 5 (7) | 3 (3) | 0 (0)
Viral (Infections and infestations) | 7 (7) | 5 (5) | 0 (0)
Allergy (General disorders) | 0 (0) | 1 (1) | 0 (0)
Device Malposition or Malfunction (Product Issues) | 1 (1) | 1 (1) | 0 (0)
Device Migration (Product Issues) | 2 (2) | 0 (0) | 0 (0)
Thrombus on Device (Product Issues) | 11 (11) | 11 (11) | 1 (1)
General-Miscellaneous (General disorders) | 87 (111) | 68 (81) | 9 (9)
Achilles Tendon Tear (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 4 (4) | 7 (7) | 0 (0)
General (Musculoskeletal and connective tissue disorders) | 7 (7) | 6 (7) | 0 (0)
General- Musculoskeletal Symptoms (Musculoskeletal and connective tissue disorders) | 12 (15) | 8 (9) | 0 (0)
General-Neurological (Nervous system disorders) | 26 (28) | 19 (19) | 1 (1)
General- Neurological Symptoms (Nervous system disorders) | 25 (26) | 13 (14) | 4 (4)
Hemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute Subdural Hematoma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
General- Opthalmologic Disorders (Eye disorders) | 3 (3) | 0 (0) | 0 (0)
General- Opthalmic Symptoms (Eye disorders) | 1 (1) | 4 (4) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0)
Chronic Obstructive Airway Disorders (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3) | 0 (0)
General- Pulmonary/Respiratory Disorders (Respiratory, thoracic and mediastinal disorders) | 27 (29) | 15 (15) | 5 (5)
Idiopathic Interstitial Lung Diseases (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural Disorders (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 13 (14) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 7 (7) | 0 (0)
X-ray Finding (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
VASC Bleeding (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 2 (2)
VASC Hematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1)
VASC Irreversible Nerve Damage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
VASC Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
VASC Pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
VASC Vessel Dissection (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
VASC Vessel Stenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/15/NCT02000115/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-25): https://cdn.clinicaltrials.gov/large-docs/15/NCT02000115/SAP_001.pdf